CLINICAL TRIAL: NCT02375178
Title: Antimicrobial Activity of Two Mouthwashes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Fernanda Sebba de Souza, student, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCAS antisseptico oral
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Periimplantitis; Dental Plaque; Periodontal Diseases; Caries; Oral Surgical Wound Infection
Keywords: anti-infective agents; local/therapeutic use; chlorhexidine; dental desinfectants; polyhexamethylene biguanide; mouthrinse
MeSH Terms: conditions — Peri-Implantitis; Dental Plaque; Periodontal Diseases | interventions — Chlorhexidine; polihexanide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sterile saline solution (Active Comparator): sterile Saline solution 0,9%
  Interventions: Drug: Sterile saline solution
- chlorhexidine (Experimental): chlorhexidine 0,12% mouthwash
  Interventions: Drug: chlorhexidine; Drug: Sterile saline solution
- polyhexamethylene (Experimental): polyhexamethylene biguanide 0,07% mouthwash
  Interventions: Drug: Polyhexamethylene biguanide; Drug: Sterile saline solution

INTERVENTIONS:
Drug: chlorhexidine — The volunteers will be instructed to mouthwash with 10ml of a sterile saline solution for 30 seconds and than make the mouthwash with 10ml of an 0.12% chlorhexidine solution. Samples of saliva will be collected immediately before the mouth wash and after 30, 60 and 180 minutes.
  Arms: chlorhexidine
Drug: Polyhexamethylene biguanide — The volunteers will be instructed to mouthwash with 10ml of a sterile saline solution for 30 seconds and than make the mouthwash with 10ml of an 0,07% solution Polyhexamethylene biguanide. Samples of saliva will be collected before the mouth wash and after 30, 60 and 180 minutes.
  Arms: polyhexamethylene
Drug: Sterile saline solution — The volunteers will be instructed to mouthwash with 10ml of a sterile saline solution for 30 seconds and than make the mouthwash with 10ml of a sterile saline solution. Samples of saliva will be collected before the mouth wash and after 30, 60 and 180 minutes.

SUMMARY:
This is a three arm randomized trial. The aim is to evaluate the antimicrobial activity of chlorhexidine and polyhexamethylene biguanide oral antiseptics on the microorganisms of the oral cavity. A total of 30 healthy volunteers will be enrolled and randomly allocated to control group (CG, n=10), which will be instructed to rinse the mouth with 10ml of a sterile saline solution for one minute, to chlorhexidine group (ClG, n=10), which will be instructed to rinse the mouth with 10ml of an 0.12% chlorhexidine solution, for one minute, or to polyhexamethylene biguanide group (PG, n=10), which will be instructed to rinse the mouth with 10ml of an 0.07% polyhexamethylene biguanide solution, for one minute. Samples of saliva will be collected before the mouth wash and after 30, 60 and 180 minutes. Samples will be plated on manitol agar, mitis salivarius agar, EMB agar and Sabouraud agar. Samples will be processed by a blinded microbiologist.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-30 years

Exclusion Criteria:

* patients with a hypersensitivity or allergic response by some component of the formula antiseptics,
* pregnant women,
* lactating,
* history of periodontal disease,
* smoking,
* decompensated diabetics,
* patients undergoing chemotherapy,
* radiotherapy patient,
* transplanted patient and refuses to participate,
* not signing a term of free and informed concentiment

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of Colony Forming Units | 180 minutes
  Samples of saliva will be collected before the mouth wash and after 30, 60 and 180 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Veiga, MD,PhD, Study Chair — Universidade do Vale do Sapucai